CLINICAL TRIAL: NCT02405858
Title: A Phase 4 Study of Zytiga in Poor-risk mCRPC (Metastatic Castration-Resistant Prostate Cancer) Patients Who Was Failed the First-line CAB (Combined Androgen Blockade) Therapy
Brief Title: A Study of Abiraterone Acetate in Metastatic Castration-Resistant Prostate Cancer Participants Who Responded Poorly to the First-line Combined Androgen Blockade Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR106841; ABI-C-14-JP-001-V03 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: Metastatic Castration-Resistant Prostate Cancer; Abiraterone Acetate; ZYTIGA; Prednisolone
MeSH Terms: interventions — Abiraterone Acetate; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Abiraterone Acetate (Experimental): Participants will receive abiraterone acetate 1000 milligram (mg) (four 250 mg tablets) orally once daily, concomitantly with oral prednisolone 10 mg per day. No food should be consumed for at least 2 hours before the dose of abiraterone acetate is taken and for at least one hour after the dose of abiraterone acetate is taken. A 28-daily dosing cycle will continue until disease progression or unacceptable toxicity is observed up to 2 years.
  Interventions: Drug: Abiraterone Acetate; Drug: Prednisolone

INTERVENTIONS:
Drug: Abiraterone Acetate — Abiraterone acetate 1000 milligram (mg) (four 250 mg tablets) orally once daily up to Cycle 26.
  Other Names: ZYTIGA
Drug: Prednisolone — Oral prednisolone 5 mg will be concomitantly administered twice a day (10 mg/day) up to Cycle 26.

SUMMARY:
The purpose of this study is to evaluate the percentage of participants achieving prostate-specific antigen (PSA) response by 12 weeks of therapy from baseline according to Prostate Cancer Clinical Trials Working Group (PCWG2) criteria.

DETAILED DESCRIPTION:
This is a Phase 4, non-randomized, multi-center (when more than one hospital work on a medical research study), open label (identity of study drug will be known to participant and study staff), single arm study of abiraterone acetate to investigate its efficacy and safety in participants with metastatic castration-resistant prostate cancer (mCRPC) who failed the first-line combined androgen blockade (CAB) therapy. The study consists of Screening Phase (28 days prior to Cycle 1 Day 1), Treatment Phase (up to 2 years), Post Treatment Phase (30 days after the last dose of study drug). Participants will receive 1000 milligram (mg) (four 250 mg tablets) of abiraterone acetate orally once daily. In addition, 5 mg of oral prednisolone will be concomitantly administered twice a day (10 mg per day). A 28-daily dosing cycle will be continued until disease progression or unacceptable toxicity is observed. The total duration of study will be 2 years. Participants will be primarily evaluated for PSA response. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have histologically or cytologically confirm adenocarcinoma of the prostate without neuroendocrine differentiation or small cell histology
* Participants who had prostate-specific antigen (PSA) progression defined as a rise of PSA at least 1 week apart resulting in 25 percent (%) increase in PSA with last PSA greater than (>) 2 nanogram per milliliter (ng/mL) (according to PCWG2) after antiandrogen withdrawal
* Participants who had PSA progression within a year after the start of first-line CAB therapy, or who had PSA progression without having a normal PSA level (less than [<] 4.0 ng/mL) in the first-line combined androgen blockade (CAB) therapy
* Participants who have not been treated with cytotoxic chemotherapy (including estramustine) for the treatment of prostate cancer (neoadjuvant or adjuvant chemotherapy is only allowed if the last dose is greater than or equal to [>=] 1 year from the scheduled date of initial administration of abiraterone acetate)
* Participants who have target or non-target metastatic abnormalities either on screening bone scan, computed tomography (CT) or magnetic resonance imaging (MRI)

Exclusion Criteria:

* A participant who has known allergies, hypersensitivity, or intolerance to abiraterone acetate or its excipients
* A participant who has severe liver dysfunction (Child-Pugh Score C), active or symptomatic viral hepatitis or chronic liver disease
* A participant who has received other hormonal therapy, including any dose of finasteride, dutasteride, any herbal product known to decrease PSA levels (example: Saw Palmetto and PC-SPES) within 4 weeks prior to the scheduled date of initial administration of abiraterone acetate
* A participant who has had surgery or local prostatic intervention within 4 weeks prior to the scheduled date of initial administration of abiraterone acetate
* A participant who has active infection or other medical condition that would make prednisolone use contraindicated

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-04-10 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Prostate-specific Antigen (PSA) Response (PSA Response Rate) by 12 Weeks of Therapy | up to 2 years
  A PSA response is defined as the first occurrence of greater than or equal to (>=) 50 percent (%) decrease from baseline by 12 weeks after the first dose of study drug, which would be subsequently confirmed by a measurement that is at least 4 or more weeks after the initial documentation.

SECONDARY OUTCOMES:
Duration of PSA Response | Up to 2 years
  Duration of PSA response was defined as the duration between the date of confirmed PSA response and subsequent PSA progression date.
Time to PSA Response | Up to 2 years
  Time to PSA response is the time from start of treatment to PSA progression.
Percentage of Participants Achieving PSA Response by 24 weeks of Therapy | Up to 2 years
  A PSA response is defined as the first occurrence of greater than or equal to (>=) 50 percent (%) decrease from baseline by 24 weeks after the first dose of study drug, which would be subsequently confirmed by a measurement that is at least 4 or more weeks after the initial documentation.
PSA-based Progression-free Survival (PSA-PFS) | Time from randomization up to radiographic progression, clinical progression or death, whichever occurs first (maximum up to 2 years)
  PSA-based Progression-free Survival is the time from randomization to the occurrence of one of the following: radiographic progression, clinical progression or death.
Maximum Serum PSA Decline Evaluation | Baseline and Day 1 of each cycle up to 2 years
  Maximum PSA Decline will be calculated as Baseline PSA level minus lowest PSA level, observed during the 2 year monthly planned PSA lab test and lowest PSA data will be used for calculating the maximum serum PSA decline.
Percentage of Participants With Radiographic Objective Response Rate (RAD-ORR) in Participants with Measurable Lesions at Baseline | Baseline, Day 1 of Cycle 1, 2,3 and 4 until first documented disease progression or up to 2 years
  Percentage of participants with radiographic objective response is defined as the percentage of participants with complete response (CR) or partial response (PR) as best overall response based on reconciled radiographic disease assessment according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.
Radiographic Progression-free Survival (RAD-PFS) | Time from enrollment up to radiographic progression or death, whichever occurs first (up to 2 years)
  RAD-PFS is defined as the time from enrollment to the occurrence of radiographic progression or death.
Time to Next Treatment | up to 2 years
  Time to next treatment was calculated as the number of days from either discontinuation of the study drug or the administration of the last dose, until the participants needed next treatment.
Overall Survival | Time from enrollment to date of death due to any cause (up to 2 years)
  Overall survival is defined as the time from enrollment to date of death due to any cause.
Brief Pain Inventory - Short Form | Baseline, Day 1 of Cycle 1, 2,3 and 4 up to 2 years
  Pain will be evaluated using the BPI-SF instrument. Total score is an average of the pain interference score (mean value for the 9 BPI-SF questions [questions inquiring about the extent of interference with activities by pain, where the extent is ranked from 0 (does not interfere) to 10 (completely interferes)]) and pain subscale score (mean value for the scores for BPI-SF questions 3, 4, 5 and 6 [questions inquiring about the extent of pain, where the extent is ranked from 0 (no pain) to 10 (pain as bad as you can imagine)]). Total score ranges from 0 to 10 with higher values indicating more pain.
Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) | up to 2 years
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; lifethreatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (14):
- Japan (14):
  - Asahi
  - Higashi-Ibaraki
  - Kanazawa
  - Kobe
  - Koshigaya
  - Kumamoto
  - Narashino
  - Okayama
  - Sagamihara
  - Sakura
  - Shinjuku-Ku
  - Sunto
  - Yokohama
  - Yokosuka

REFERENCES:
- See also: A Phase 4 Study of Abiraterone Acetate in Metastatic Castration-Resistant Prostate Cancer Patients Who Poorly Responded to the First-line Combined Androgen Blockade Therapy — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR106841&attachmentIdentifier=79e26442-4a50-4f25-82f6-4c35ae397eed&fileName=CR106841_CSR.pdf&versionIdentifier=